CLINICAL TRIAL: NCT03298113
Title: Effects of an Advanced Skin Protectant in the Management of Incontinence-associated Dermatitis Compared to Hospital Standard Care Practice: an Exploratory Randomized Controlled Trial
Brief Title: Comparative Study to Assess an Advanced Skin Protectant in the Management of Incontinence-associated Dermatitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow enrollment
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLIN-PROT-EU-05-293312
Record Dates: First submitted 2017-08-21; First posted 2017-10-02 (Actual); Results first posted 2019-09-24 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Incontinence-associated Dermatitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Central reader
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Cavilon Advanced Skin Protectant (Experimental): Product applicator contains liquid barrier and is applied according to the 3M manufacturer's instructions for use.
  Interventions: Device: Cavilon Advanced Skin Protectant
- IAD Hospital Standard Care (Other): Marketed products are applied according to the IAD hospital standard care routine.
  Interventions: Device: IAD Hospital Standard Care

INTERVENTIONS:
Device: Cavilon Advanced Skin Protectant — Applicator contains a polymeric-cyanoacrylate solution intended to cover and protect intact or damaged skin. Upon application to skin, the liquid dries rapidly to form a primary long-lasting waterproof, highly durable film barrier.
  Arms: Cavilon Advanced Skin Protectant
Device: IAD Hospital Standard Care — Devices such as local skin protectants will be used according to the hospital IAD care regime and under consideration of the respective manufacturers' instructions for use.
  Arms: IAD Hospital Standard Care

SUMMARY:
The purpose of the clinical study is to assess the effects of 3M Cavilon Advanced Skin Protectant in comparison to different local IAD care regimes in hospitals (IAD: Incontinence-associated Dermatitis)

DETAILED DESCRIPTION:
The purpose of the clinical study is to assess the effects of 3M Cavilon Advanced Skin Protectant in comparison to different local IAD care regimes in hospitals (IAD: incontinence-associated dermatitis). IAD is a skin damage caused by exposure to moisture and irritants such as urine and/or stool. The clinical appearance ranges from painful erythema to severe erosion and denudation/skin loss with or without secondary infection. The durable, long lasting skin protectant (3M study device) is formulated to attach to moist or wet skin surfaces (i.e., superficial, partial thickness skin loss) to provide better protection against moisture and irritants under challenging conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Is the patient 18 years or older?
2. Has the patient or their legally authorized representative signed the Informed Consent Form?
3. Does the patient have IAD category 1A (IAD 1A: persistent redness without clinical signs of infection) or IAD category 2A (IAD 2A: skin loss without clinical signs of infection) in the study area (study area: the sacral region going down to the upper thighs, bordered approximately 5 cm below the gluteal fold?
4. Is the patient incontinent and does stool and/or urine come into direct contact with the skin?
5. Is the patient able to be turned/positioned with regard to skin assessment and photo documentation?
6. Is there a reasonable expectation that the patient will remain in the hospital setting for at least 7 days?

Exclusion Criteria:

1. Is the patient pregnant or breast feeding?
2. Does the patient have a known hypersensitivity or allergy to acrylate or cyanoacrylate?
3. Does the patient have a stage II, III, IV or unstageable pressure ulcer or other suspected deep tissue injury in the study area?
4. Does the patient require topical treatment due to a fungal, bacterial or viral infection in the study area?
5. Does the patient require treatment with topical medication or product other than IAD treatment in the study area?
6. Does the patient have any other local dermatological disease or skin condition interfering with this study?
7. Does the patient have any medical condition (e.g. end of life, planned elective surgery) that in the opinion of the investigator should exclude him/her from participating in the study?
8. Does the patient participate in another study with a known or implied effect on skin barrier function?

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew M. Cooper, MD, Study Director — 3M
Locations (3):
- Universitair Ziekenhuis Gent, Ghent, East Flanders, Belgium
- Charité - Universitätsmedizin Berlin, Berlin, Germany
- University Hospital Southampton, Southampton, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cavilon Advanced Skin Protectant | IAD Hospital Standard Care
Started | 10 (10 subjects were treated w/ Cavilon Advanced Skin Protectant. Study terminated due to low enrollment) | 10 (10 subjects were treated with IAD Hospital Standard Care. Study terminated due to low enrollment.)
IAD 1A | 3 | 4
IAD 2A | 7 | 6
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients with Incontinence-associated Dermatitis
Groups:
- Total: Total of all reporting groups
Arm/Group | Cavilon Advanced Skin Protectant | IAD Hospital Standard Care | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 8 | 10 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 2 | 5 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Belgium | 4 | 4 | 8
  Germany | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Healing of IAD
Description: Number and percentage of patients completely healed (skin free of any IAD signs, including erythema, based on a structured skin assessment according to the GLOBIAD criteria (GLOBIAD: Ghent Global IAD Categorization Tool)
  Note: Due to the exploratory design no formal a priori hypothesis was defined for this study. The outcome measure type for all endpoints is "other pre-specified". The effects were analyzed using descriptive statistics. No confirmatory statements can be made about the effects and no comparative statements are possible. The sponsor decided to early terminate the study after 20 evaluable patients for the intention-to-treat analysis. Reason for the early termination was the slow enrollment rate of patients and overall short length of stay in hospital.
Time Frame: up to 21 days depending on length of hospitalization
Population: Analysis was done based on the intention-to-treat (ITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Cavilon Advanced Skin Protectant | IAD Hospital Standard Care
Number analyzed (Participants) | 10 | 10
Participants
  Not completely healed | 10 | 9
  Completely healed | 0 | 1

2. Other Pre Specified Outcome: Improvement of IAD Category
Description: Number and percentage of patients improved with regard to IAD category
Time Frame: Up to 21 days depending on length of hospitalization
Population: Analysis was done based on the intention-to-treat (ITT) population. In both treatment groups, there were two improvements in the IAD category for patients who started with IAD 2A (IAD 2A: skin loss without clinical signs of infection) and switched to IAD 1A (IAD 1A: persistent redness without clinical signs of infection).
Measure: Count of Participants; unit: Participants
Arm/Group | Cavilon Advanced Skin Protectant | IAD Hospital Standard Care
Number analyzed (Participants) | 10 | 10
Participants
  Worsened | 0 | 0
  Remained the Same | 8 | 8
  Improved | 2 | 2

3. Other Pre Specified Outcome: Re-epithelialization of Skin Loss
Description: Number and percentage of patients with 100% re-epithelialization of skin loss based on structured skin assessment (skin loss: skin is moist, as the epidermal layer is missing).
Time Frame: up to 21 days depending on length of hospitalization
Population: Analysis was done based on the IAD 2A patient population at start of study (IAD 2A: skin loss without clinical signs of infection)
Measure: Count of Participants; unit: Participants
Arm/Group | Cavilon Advanced Skin Protectant | IAD Hospital Standard Care
Number analyzed (Participants) | 7 | 6
Participants
  Not completely ephitelialized | 5 | 4
  Completely epithelialized | 2 | 2

4. Other Pre Specified Outcome: Time to Heal IAD
Description: Time to complete healing of IAD in the terms of days of treatment (skin free of any IAD signs, including erythema, based on a structured skin assessment according to the GLOBIAD criteria (GLOBIAD: Ghent Global IAD Categorization Tool)
Time Frame: Up to 21 days depending on length of hospitalization
Population: Analysis was done based on the intention-to-treat (ITT) population. No healing event occured in the arm/group treated with Cavilon Advanced Skin Protectant in this study.
Measure: Number; unit: Days
Units Other Than Participants: Healing Events
Arm/Group | Cavilon Advanced Skin Protectant | IAD Hospital Standard Care
Number analyzed (Participants) | 10 | 10
Number analyzed (Healing Events) | 0 | 1
Days |  | 13.00

5. Other Pre Specified Outcome: Time to Improve in IAD Category
Description: Time to improve in IAD category in the terms of days of treatment.
Time Frame: Up to 21 days depending on length of hospitalization
Population: Analysis was done based on the intention-to-treat (ITT) population. In both treatment groups, there were two improvements in the IAD category for patients who started with IAD 2A (skin loss without clinical signs of infection) and switched to IAD 1A (persistent redness without clinical signs of infection).
Measure: Mean (Standard Deviation); unit: Days
Units Other Than Participants: Improvement Events
Arm/Group | Cavilon Advanced Skin Protectant | IAD Hospital Standard Care
Number analyzed (Participants) | 10 | 10
Number analyzed (Improvement Events) | 2 | 2
Days | 9.50 (0.707) | 5.50 (2.121)

6. Other Pre Specified Outcome: Prevention of Skin Loss
Description: Protection of IAD category 1 patients from developing IAD category 2
Time Frame: up to 21 days depending on length of hospitalization
Population: Analysis was done based on the IAD 1A patient population at start of study (IAD 1A: persistent redness without clinical signs of infection)
Measure: Count of Participants; unit: Participants
Arm/Group | Cavilon Advanced Skin Protectant | IAD Hospital Standard Care
Number analyzed (Participants) | 3 | 4
Participants
  Worsened | 0 | 0
  Remained the Same | 3 | 4
  Improved | 0 | 0

7. Other Pre Specified Outcome: Prevention of IAD Recurrence
Description: Protection of completely healed patients from recurrence of IAD during the study.
Time Frame: up to 21 days depending on length of hospitalization
Population: The overall number of participants analyzed represents the number of patients completely healed during this study.
  No healing event occured in the group treated with Cavilon Advanced Skin Protectant and therefore prevention of IAD recurrence could no be assessed. One healing event occured in the group treated with IAD Hospital Standard Care.
Measure: Number; unit: IAD Recurrence Events
Arm/Group | Cavilon Advanced Skin Protectant | IAD Hospital Standard Care
Number analyzed (Participants) | 0 | 1
IAD Recurrence Events |  | 0

8. Other Pre Specified Outcome: Product Cost: IAD 1A
Description: Mean average daily product cost per patient for IAD 1A treatment based on skin protectant utilization such as type of skin protectant, frequency of application and days of treatment.
  Note: One patient in the group treated with Cavilon Advanced Skin Protectant stayed only one day in the study due to an unrelated Severe Adverse Event at night. This had an impact on the product cost calculation. The application interval for Cavilon Advanced Skin Protectant in this study was three days (D1, D4, D7, D10, D13, D16, D19) , while the use of IAD products for standard hospital care was based on manufacturer recommendations, which could correspond to a daily interval with multiple applications.
Time Frame: up to 21 days depending on length of hospitalization
Population: Analysis was done based on the IAD 1A population at start of study (IAD1A: persistent redness without clinical signs of infection).
Measure: Mean (Standard Deviation); unit: Euro
Arm/Group | Cavilon Advanced Skin Protectant | IAD Hospital Standard Care
Number analyzed (Participants) | 3 | 4
Euro | 5.56 (3.80) | 0.75 (0.06)

9. Other Pre Specified Outcome: Product Cost : IAD 2A
Description: Mean average daily cost per patient for IAD 2A treatment based on skin protectant utilization such as type of skin protectant, frequency of application and days of treatment
Time Frame: up to 21 days depending on length of hospitalization
Population: Analysis was done based on the IAD 2A population at start of study (IAD 2A: Skin loss without clinical signs of infection)
Measure: Mean (Standard Deviation); unit: Euro
Arm/Group | Cavilon Advanced Skin Protectant | IAD Hospital Standard Care
Number analyzed (Participants) | 7 | 6
Euro | 4.67 (2.53) | 1.21 (1.34)

10. Other Pre Specified Outcome: Use of Resources Involved in IAD Therapy
Description: Additional appointments with specialists involved in IAD therapy
Time Frame: Up to 21 days depending on length of hospitalization
Population: Analysis was done based on the intention-to-treat (ITT) population
Measure: Number; unit: Appointments
Arm/Group | Cavilon Advanced Skin Protectant | IAD Hospital Standard Care
Number analyzed (Participants) | 10 | 10
Appointments | 0 | 0

11. Other Pre Specified Outcome: Nursing Time Related to Cleansing
Description: Nursing time to clean up incontinence episode
Time Frame: up to 21 days depending on length of hospitalization
Population: Analysis was done based on the intention-to-treat (ITT) population Note: One patient allocated to Cavilon Advanced Skin Protectant participated in the study for only one day. Therefore, the time required to clean up the incontinence episode could not be measured (n = 1 missing data set; only 9 data sets were available for analysis).
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Cavilon Advanced Skin Protectant | IAD Hospital Standard Care
Number analyzed (Participants) | 9 | 10
Minutes | 13.67 (7.99) | 12.41 (8.17)

12. Other Pre Specified Outcome: Nursing Time Related to Product Application
Description: Nursing time to administer skin protectants for IAD treatment
Time Frame: up to 21 days depending on length of hospitalization
Population: Analysis was done based on the intention-to-treat (ITT) population Note: For two patients allocated to Cavilon Advanced Skin Protectant the nursing time to administer the skin protectant was not recorded (n = 2 missing data sets; only 8 data sets were available for analysis).
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Cavilon Advanced Skin Protectant | IAD Hospital Standard Care
Number analyzed (Participants) | 8 | 10
Minutes | 2.49 (3.20) | 2.02 (1.90)

13. Other Pre Specified Outcome: Pain Related to Cleansing: IAD 1A
Description: Pain scores related to clean up incontinence episode for IAD 1A patients. The table details the reduction in pain experienced by subjects able to report their last recorded cleaning event relative to baseline. More extreme negative values denote a larger reduction in pain. For cleansing, IAD 1A patients treated with Cavilon Advanced Skin Protectant saw no change in pain due to having no pain reported at baseline nor last visit.
  Note: For this study the Wong-Baker FACES® Pain Rating Scale was used for patients able to report pain. Faces with different expressions from smiling to crying facilitated the communication as anchor for pain intensity scale (scores: 0, 2, 4, 6, 8, 10), with higher score indicating more pain.
Time Frame: up to 21 days depending on length of hospitalization
Population: Analysis was done based on the IAD 1A study population at start of study (IAD 1A: persistent redness without clinical signs of infection) Note: One patient allocated to IAD Hospital Standard Care was not able to report pain (n = 1 missing data set; only n = 3 data sets were available for analysis)
Measure: Mean (Standard Deviation); unit: Change in score on a scale
Arm/Group | Cavilon Advanced Skin Protectant | IAD Hospital Standard Care
Number analyzed (Participants) | 3 | 3
Change in score on a scale | 0.00 (0.000) | -2.00 (3.464)

14. Other Pre Specified Outcome: Pain Related to Cleansing: IAD 2A
Description: Pain scores related to clean up incontinence episode for IAD 2A patients. The table details the reduction in pain experienced by subjects able to report their last recorded cleaning event relative to baseline. More extreme negative values denote a larger reduction in pain.
  Note: For this study the Wong-Baker FACES® Pain Rating Scale was used for patient able to report pain. Faces with different expressions from smiling to crying facilitated the communication as anchor for pain intensity scale (scores: 0, 2 , 4, 6, 8, 10), with higher score indicating more pain.
Time Frame: up to 21 days depending on length of hospitalization
Population: Analysis was done based on the IAD 2A population at start of study (IAD 2A: skin loss without clinical signs of infection) Note: One patient allocated to Cavilon Advanced Skin Protectant was not able to report pain (n = 1 missing data set; only n = 6 data sets were available for analysis)
Measure: Mean (Standard Deviation); unit: Change in score on a scale
Arm/Group | Cavilon Advanced Skin Protectant | IAD Hospital Standard Care
Number analyzed (Participants) | 6 | 6
Change in score on a scale | -3.00 (4.147) | -0.33 (4.274)

15. Other Pre Specified Outcome: Pain Related to Product Application: IAD 1A
Description: Pain scores related to application of skin protectants for IAD 1A patients (Wong-Baker FACES® Pain Rating Scale). The table details the reduction in pain experienced by subjects able to report at their last recorded application event relative to baseline.
  Note: For this study the Wong-Baker FACES® Pain Rating Scale was used for patient able to report pain. Faces with different expressions from smiling to crying facilitated the communication as anchor for pain intensity scale (scores: 0, 2 , 4, 6, 8, 10), with higher score indicating more pain.
Time Frame: up to 21 days depending on length of hospitalization
Population: Analysis was done based on the IAD 1A population at start of study (IAD 1A: persistent redness without clinical signs of infection) Note: One patient allocated to IAD Hospital Standard Care was not able to report pain (n = 1 missing data set, only n= 3 data sets were available for analysis)
Measure: Mean (Standard Deviation); unit: Change in score on a scale
Arm/Group | Cavilon Advanced Skin Protectant | IAD Hospital Standard Care
Number analyzed (Participants) | 3 | 3
Change in score on a scale | 0.00 (0.000) | 0.00 (0.000)

16. Other Pre Specified Outcome: Pain Related to Product Application: IAD 2A
Description: Pain scores related to application of skin protectants for IAD 2A patients (Wong-Baker FACES® Pain Rating Scale). The table details the reduction in pain experienced by subjects able to report at their last recorded application event relative to baseline. More extreme negative values denote a larger reduction in pain.
  Note: For this study the Wong-Baker FACES® Pain Rating Scale was used for patient able to report pain. Faces with different expressions from smiling to crying facilitated the communication as anchor for pain intensity scale (scores: 0, 2 , 4, 6, 8, 10), with higher score indicating more pain.
Time Frame: up to 21 days depending on length of hospitalization
Population: Analysis was done based on IAD 2A population at start of study (IAD 2A: skin loss without clinical signs of infection) Note: One patient in the Cavilon Advanced Skin Protectant group and one patient in the IAD Hospital Standard care group were not able to report pain.
Measure: Mean (Standard Deviation); unit: Change in score on a scale
Arm/Group | Cavilon Advanced Skin Protectant | IAD Hospital Standard Care
Number analyzed (Participants) | 6 | 5
Change in score on a scale | -2.33 (4.082) | -1.20 (5.020)

ADVERSE EVENTS:
Time Frame: 9 months
Description: ISO 14155 Definitions (ISO: International Organization for Standardization)
Arm/Group | Cavilon Advanced Skin Protectant | IAD Hospital Standard Care
All-Cause Mortality (participants affected / at risk) | 0/10 | 1/10
Serious Adverse Events (participants affected / at risk) | 1/10 | 1/10
Other Adverse Events (participants affected / at risk) | 6/10 | 2/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cavilon Advanced Skin Protectant (N=10) | IAD Hospital Standard Care (N=10)
Cardiac arrest (Cardiac disorders) | 1 | 0
Acute renal failure (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cavilon Advanced Skin Protectant (N=10) | IAD Hospital Standard Care (N=10)
Fungal infection (Infections and infestations) | 2 | 2
Clostridium difficile infection (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 0
Device adhesion issue (Product Issues) | 1 | 0
Vaginal mycosis (Infections and infestations) | 1 | 0

LIMITATIONS AND CAVEATS:
Early termination due to slow enrollment rate and overall short length of hospital stay leading to small numbers of subjects analyzed (n = 20 ITT). No confirmatory and comparative statements can be made about the effects (exploratory study design).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/13/NCT03298113/Prot_SAP_000.pdf